CLINICAL TRIAL: NCT06240442
Title: Bodyweight Interval Exercise in the Fed Versus Fasted State on Postprandial Glycemia, Appetite Perceptions and Fat Oxidation
Brief Title: Bodyweight Interval Exercise in the Fed Versus Fasted State
Acronym: BWE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Jenna Gillen, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 40799
Record Dates: First submitted 2024-01-14; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasted Exercise (Experimental): Exercise followed by breakfast
  Interventions: Other: Fasted exercise
- Fed Exercise (Experimental): Breakfast followed by exercise
  Interventions: Other: Fed exercise

INTERVENTIONS:
Other: Fasted exercise — Bodyweight interval exercise performed 5 minutes before the start of a mixed-macronutrient breakfast meal
  Arms: Fasted Exercise
Other: Fed exercise — Bodyweight interval exercise performed 10 minutes after the start of consuming a mixed-macronutrient breakfast meal
  Arms: Fed Exercise

SUMMARY:
The purpose of this study is to investigate the effects of a single session of at-home bodyweight interval exercise, performed in the fasted or fed state, on postprandial glycemic management, post-exercise fat oxidation, and overall perceptions of appetite in recreationally active females. This is a remote/online study and does not involve any visits to the laboratory.

DETAILED DESCRIPTION:
Following the acquisition of informed consent via videoconferencing, eligibility to participate in the study will be determined using questionnaires. If inclusion criteria is met, participants will undergo virtual exercise familiarization by following a pre-recorded instructional video.

Eligible participants will be assigned, in a random order, to two metabolic trials at least 3 days apart in the follicular phase of the same menstrual cycle. These visits will be online with an investigator on videoconferencing. The two trials involve: 1) Exercise followed by breakfast; and 2) Breakfast followed by exercise.

Various outcomes will be measured throughout the metabolic trials including: blood sugar, fat oxidation and appetite. All research tools needed to acquire these methods will be delivered to participants' place of residence.

ELIGIBILITY:
Inclusion Criteria:

* Females 18-35 years
* Recreationally active (complete <150 min of exercise 1-3 days per week) and not training for any specific sport
* Experiencing monthly menstrual periods (eumenorrheic)
* Are not currently on oral contraceptives, or are taking triphasic oral contraceptives
* Body mass index (BMI) ≥18.5 kg/m2 and ≤30 kg/m2
* Regular consumption of a breakfast meal (solid and liquid meals apply) most (≥ 4) days of the week
* Have a device compatible for use with study applications (e.g., smart phone)

Exclusion Criteria:

* Inability to safely perform physical activity as determined by the Get Active Questionnaire
* Not willing to consume the standardized test drink before and after exercise
* Sensitive to meal timing around exercise (e.g., gastrointestinal issues if exercise performed 10 min after the start of meal consumption or if a meal is consumed 5 min after exercise)
* Inability to adhere to pre-trial protocol guidelines (e.g., caffeine or alcohol restrictions)
* Physical limitations for bodyweight exercise
* Are on monophasic or biphasic oral contraceptives
* Regular tobacco or cannabis use (e.g., recreational and/or medical cannabis, cigarettes, e-cigarettes, vape pens, JUUL)
* Regular use of drugs that may alter metabolism (e.g., corticosteroids, nSAIDs)
* Diagnosed medical condition under the care of care of a physician (e.g., type 2 diabetes, cardiovascular disease) Currently enrolled in a course with Dr. Gillen

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Average blood glucose concentration | 2 hours
  Average blood glucose concentration during postprandial period

SECONDARY OUTCOMES:
Blood glucose concentration | 2 hours
  Blood glucose concentration across postprandial period
Blood glucose area under the curve | 2 hours
  blood glucose area under the curve during postprandial period
Peak blood glucose concentration | 2 hours
  peak glucose across postprandial period
Post-exercise fat oxidation | pre-exercise, immediately post-exercise, up to 3 hours post-exercise
  post-exercise fat oxidation measured as percent carbon dioxide
Appetite Perceptions | pre-exercise, immediately post-exercise, and 1, 2 and 3 hours post-exercise
  Visual analog scales (0-100) will be used to determine perceptions of hunger, satisfaction, fullness, and prospective food consumption with higher scores denoting increased perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Gillen, PhD, Principal Investigator — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No